CLINICAL TRIAL: NCT01133353
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Tetrabenazine MR in Subjects Aged 5 up to 17 Years With Tourette's Syndrome
Brief Title: A Study of the Effectiveness and Safety of Tetrabenazine MR in Pediatric Subjects With Tourette's Syndrome
Acronym: TBZ-MR
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BVF-018-201
Record Dates: First submitted 2010-05-24; First posted 2010-05-28 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Tourette's Syndrome
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tetrabenazine MR (Experimental)
  Interventions: Drug: Tetrabenazine MR
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tetrabenazine MR — Modified-Release (MR) tablets containing 15 mg or 30 mg tetrabenazine, dose-escalating up to a maximum of 150 mg depending on weight, once per day for 12 weeks
  Arms: Tetrabenazine MR
Drug: Placebo — 1 to 5 tablets once per day depending on weight for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to study the therapeutic effect of tetrabenazine MR in children with Tourette's Syndrome, as measured by the improvement in total tic score of the Yale Global Tic Severity Scale (YGTSS).

DETAILED DESCRIPTION:
Tourette's Syndrome (TS) is typically diagnosed in early childhood (6-7 years) or before the age of 21 years and is characterized by chronic, intermittent motor and phonic tics. There is a body of evidence, mostly from the clinical experience data, suggesting the efficacy of tetrabenazine in TS patients with tics, including patients who were unresponsive to other treatment options. These publications consistently report the usefulness of tetrabenazine as an alternative to conventional neuroleptics for the treatment of TS.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria:

1. Children aged 5 to up to 17 years
2. Subjects must be capable of providing informed consent or assent, if applicable, and parents/legal guardian must be capable of providing informed consent/permission and complying with study procedures
3. Subject and parents/legal guardian must be able to communicate effectively with Investigator and study coordinator
4. Diagnosed with Tourette's Syndrome, according to DSM-IV-TR and using K-SADS-PL to aid diagnosis, and requiring drug therapy
5. Total tic score ≥ 22 as measured by YGTSS at screening and baseline
6. Total body weight ≥ 15 kg (33 lbs.)
7. Tics are causing distress or impairment, as determined by parent/legal guardian or subject and by the Investigator, despite current treatment regimen
8. Able to swallow whole tablets without difficulty
9. Non-pregnant status:

   * All female subjects must be non-pregnant (as demonstrated by negative serum β-HCG test), non-breastfeeding, and must avoid pregnancy from at least 10 days before signing the informed consent/assent and up until 1 month after the end of the study by abstaining from sexual activity or using two (2) medically acceptable methods of contraception, such as: a non-hormonal IUD with spermicide, female condom with spermicide, contraceptive sponge with spermicide, an intravaginal system, diaphragm with spermicide, cervical cap with spermicide, a male sexual partner who agrees to use a male condom with spermicide, a sterile sexual partner.
   * Male subjects must abstain from sexual activity from the time they sign the informed consent/assent and up until 1 month after the end of the study or use a condom with spermicide.
   * For all females of child bearing potential, a serum pregnancy test result must be negative at Screening and urine pregnancy test must be negative at Baseline

Exclusion Criteria:

Subjects are not eligible if any of the following criteria are met:

1. Subjects with history or current major depressive disorder
2. Prior treatment with > 7 doses of tetrabenazine
3. Prior treatment with reserpine
4. Subjects with impaired renal function (defined as having a creatinine level of ≥ 1.5 times the upper limit of age-appropriate normal value)
5. Subjects with current or any history of suicidal ideation
6. Participation in an investigational medication trial within the 3 months prior to the Screening visit, except for study BVF-018-102
7. Use of Botox® (botulinum toxin) within the 4 months prior to the Screening visit
8. Immediate families of site Investigators or sponsor employees
9. Excluding conditions related directly to the disease under study, subject has a history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or oncologic or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
10. Subjects with clinically important thyroid dysfunction requiring medication
11. Subjects with impaired hepatic function (defined as having SGOT/SGPT levels ≥ 1.5 times the upper limit of age-appropriate normal values)
12. Subjects with a Children's Depression Rating Scale-Revised (CDRS-R) total score of > 65
13. Male subjects with QTc > 450 msec; female subjects with QTc > 470 msec based on Bazzett's correction formula
14. Organic brain disease, for example, traumatic brain injury residua or toxic delirium
15. Any subject at immediate risk of requiring hospitalization
16. Physical examination, electrocardiography, or laboratory values that are clinically important in the opinion of the Investigator
17. Autistic spectrum disorder
18. Schizophrenia
19. Other psychotic disorder
20. Subjects with Bipolar I Disorder
21. Subjects with one or more first-degree relatives with Bipolar I Disorder
22. Subjects who are unable to complete a washout period of 4 weeks for fluoxetine and 3 weeks for MAOIs, respectively, prior to Baseline visit and who require fluoxetine and MAOIs during the Treatment Period
23. Inability to washout of strong inhibitors or inducers of CYP2D6 within 7 days of the Baseline visit
24. Positive findings on urine drug screen at the Screening Visit
25. Allergies to tetrabenazine or its excipients

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in total tic score as measured by the Yale Global Tic Severity Score (YGTSS) | Days 0 to 84

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of tetrabenazine using cognitive measures | Days 0 and 84
To evaluate the safety and tolerability of tetrabenazine using an assessment of depression | Days 0 to 84
To evaluate the safety and tolerability of tetrabenazine using an assessment of suicidality | Days 0 to 91
To explore the therapeutic effects of tetrabenazine using the full YGTSS | Days 0 to 84
To explore the therapeutic effects of tetrabenazine using the Patient Global Impression of Change scale (PGI-C) | Days 0 to 84
To explore the therapeutic effects of tetrabenazine using the Clinical Global Impression of Severity scale (CGI-S) | Days 0 to 84